CLINICAL TRIAL: NCT07049861
Title: Increasing Access to USPSTF-Recommended Obesity Care for Youth and Adults Who Are Recipients of Medicaid: Evaluation of a Comprehensive Multidisciplinary Obesity Care Training Program in FQHCs
Brief Title: Advancing Biopsychosocial Care Training Initiative
Acronym: ABC Initiative
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); Children's Mercy Hospital Kansas City (Other); University of Missouri-Columbia (Other); Missouri Institute of Mental Health (Unknown); University of Missouri, Kansas City (Other); The Missouri Department of Social Services, MO HealthNet Division, Office of Transformation (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 202406146; 5R01DK134961 (NIH)
Record Dates: First submitted 2025-06-25; First posted 2025-07-03 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-12

CONDITIONS: Weight Management; Obesity Prevention; Obesity and Obesity-related Medical Conditions; Obesity and Overweight; Obesity
Keywords: Training; Implementation; Intensive Behavioral Treatment; Family-based Behavioral Treatment; Obesity; Obesity Care
MeSH Terms: conditions — Obesity; Overweight

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CMOC (Active Comparator): The Provider Trainees at the Federally Qualified Health Centers (FQHCs) assigned to the Comprehensive Multidisciplinary Obesity Care (CMOC) condition will receive the CMOC Training during the12-month training period (months 0-12) of the trial, followed by a 12-month (month 13-24) sustainability period.
  Interventions: Other: Comprehensive Multidisciplinary Obesity Care
- IAUC (Active Comparator): The Provider Trainees at the Federally Qualified Health Centers (FQHCs) in the implementation as usual control (IAUC) condition will receive the IAUC Training during the12-month training period (months 0-12) of the trial, followed by a 12-month (month 13-24) sustainability period. Following the 12-month sustainability period, Provider Trainees will be offered the CMOC Training.
  Interventions: Other: Comprehensive Multidisciplinary Obesity Care; Other: Implementation as Usual Control

INTERVENTIONS:
Other: Comprehensive Multidisciplinary Obesity Care — CMOC is an innovative approach to obesity care delivery that leverages policy, clinical and community linkages, and digital technology for scalability. CMOC involves training providers (medical providers, registered dietitians, and behavioral health providers) to deliver guideline-based obesity care for youth and adults with obesity who receive Medicaid. Guidelines-based care involves screening, identification, weight counseling, and referral to intensive behavioral treatment by medical providers, and delivery of multicomponent intensive behavioral treatment by behavioral health providers and registered dietitians.
  Other Names: Core+
Other: Implementation as Usual Control — The standard of care implemented in FQHCs in the absence of CMOC training.
  Other Names: Core
  Arms: IAUC

SUMMARY:
This project will compare two training approaches for US Preventive Services Task Force recommended obesity care in Federally Qualified Health Centers (FQHC) across four aims. Aim 1 compares patient-level effectiveness [i.e., patient relative weight change and the proportion of patients who achieve clinically significant weight loss]. Aim 2 compares reach (patient treatment utilization). Aim 3 compares primary care provider (PCP) referrals to USPSTF-recommended care at 12 (adoption) and 24 months (maintenance) and short- and long-term changes in provider obesity care competencies . Aim 4 compares implementation and service costs.

ELIGIBILITY:
Study Eligibility Criteria - Provider Trainees:

* Provider Trainees must be PCPs, BHPs, RDNs, or CHWs who work at participating clinics.

  * PCPs that are eligible to participate as Provider Trainees can be any of the following: Medical Doctors (MD), Doctor of Osteopathic Medicine (DO), Physician Assistants (PA), or Nurse Practitioners (NP). PCPs must see patients in a primary care setting and be capable of referring patients to IBT and MNT. PCPs must have already completed their residency (when applicable).
  * BHPs that are eligible to participate as Provider Trainees must be at least one of the following categories (listed with typical credentials): Licensed Clinical Social Worker (LCSW), Licensed Professional Counselor (LPC), Licensed Marriage and Family Therapist (LMFT), Psychologist (PhD/PsyD), Psychiatric Nurse Practitioner, Psychiatrist (MD).
  * RDNs that are eligible to participate as Provider Trainees must be Registered Dietitians/Registered Dietitian Nutritionists.
  * CHWs must work as Community Health Workers, or in functionally similar role, within participating clinics

Study Eligibility - EHR Patients: Benefit-Eligible Patients from Participating Clinics

* Benefit-Eligible Patients from Participating Clinics can either be youth (ages 5-20) or adults (ages 21+) and must be recipients of Medicaid, eligible for the MO Medicaid benefit (i.e., Medicaid recipients with obesity), and have been seen at participating FQHC clinics.

Exclusion Criteria - Provider Trainees:

* Not at a participating clinic
* PCPs who do not have the ability to refer to IBT or MNT
* Resident Doctors
* A doctor specializing in reproductive health (or related fields)

Exclusion Criteria - Benefit-Eligible Patients from Participating Clinics:

* Patients without obesity
* Patients not on Medicaid
* Youth under the age of 5
* Not a patient at a participating clinic

Min Age: 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 6200 (Estimated)
Dates: Start 2025-07-09 (Actual); Primary Completion 2029-07-31 (Estimated); Study Completion 2029-07-31 (Estimated)

PRIMARY OUTCOMES:
Change in patient percent overweight | Months 2-29 post-enrollment
  Percent over the median body mass index (BMI) for sex and age.

CONTACTS AND LOCATIONS:
Overall Officials: Denise Wilfley, Ph.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu